CLINICAL TRIAL: NCT06100094
Title: Qualitative Study on CRIAVS-LR (Resource Centre for Sex Offenders in Languedoc-Roussillon, France) Psychoeducation Group for Juvenile Sex Offenders
Brief Title: Qualitative Study on a Psychoeducation Group for Juvenile Sex Offenders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-MTP_2023_09_202301455
Record Dates: First submitted 2023-10-10; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Sex Offense
Keywords: juvenile sex offenders; support group; psychoeducation; paraphilia; pedophilic interest; sexual violence
MeSH Terms: conditions — Paraphilic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- juvenile sex offender psychoeducation group: The psychoeducation group consists of 10 sessions of approximately 1.5 hours each, once a week or every two weeks depending on the availability of the therapists. Among the sessions, 9 correspond to a specific theme: reminder of the law and violence, sexism, consent, control, social pressure, self-control, empathy, seduction and romantic relationships, sex under the influence. The last session is devoted to a resumption of all the themes previously discussed. Semi-structured qualitative interviews addressing their feelings regarding the psychoeducation group, what they learned from it, what they had difficulty with.
  Interventions: Other: semi-structured qualitative interviews

INTERVENTIONS:
Other: semi-structured qualitative interviews — During the interview, a list of semi-open questions will be asked :
  * What were your expectations/state of mind before the group?
  * How would you describe your experience overall?
  * If you had to describe the group how would you do it?
  * Between two group sessions, how did it go for you?
  * What do you think of the group ultimately?
  Interviews will be carried out until data saturation.
  Collection of socio-demographic data (age), medical history and criminal history in the patient's file

SUMMARY:
Some sexual violence is committed by minors but how to take care of them ? Despite heterogeneous profiles, some characteristics are common in these adolescents and can be used in psychoeducation group. CRIAVS-LR team has therefore decided to create a psychoeducation group on emotional and sexual life specific for this population of young adult/adolescents in order to improve their skills and find alternative solutions to violence, particularly in the area of sexual violence The qualitative aspect of this study would make it possible to provide data in this still little explored field, to try to understand the experience of the young people participating in this group and to improve its structure and content so that it reaches best its goals.

DETAILED DESCRIPTION:
In France, 25% of perpetrators of sexual offenses are minors. Faced with this increasingly present problem in our society, the answer seems to be more on the side of education and care. However, this new problem confronts us with the limits of our care and forces us to reconsider the organization of care. Indeed, to date, there is no specific support for juvenile sex offenders. Little research exists on the subject because of the many difficulties in setting up this type of study: low power, problem of definition, variables that are difficult to compare, few therapists specialized in this field... In fact, studies must continue to demonstrate the effectiveness of psychoeducational treatment. Although there is no consensus on the profiles of juvenile sex offenders in the literature, there are common characteristics among these individuals. Indeed, the lack of social skills, relationship difficulties, empathy, self-esteem, sex education, impulse control and therefore self-control are issues that can be worked on by psychoeducation.

CRIAVS-LR's team have therefore decided to create a specific psychoeducation group for minors and young adults who are perpetrators of sexual violence. The objective is to improve their skills of knowing, knowing how to be and knowing how to do in the areas of affective and sexual interpersonal relationships and thus find alternative solutions to violence, particularly sexual violence. The qualitative aspect of this study would make it possible to provide data in this still little explored field, to try to understand the experience of the young people participating in this group and to improve its structure and content so that it reaches best its goals.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 14 to 20
* commit a sexual offense
* takes part to CRIAVS-LR psychoeducation group

Exclusion Criteria:

* severe intellectual disability, decompensated psychiatric disease
* Illiterate or unable to understand the purpose and methodology of the study
* Patient not affiliated to a French social security scheme or not a beneficiary of such a scheme
* Person unable to give consent
* Refusal of consent after information
* Adult protected by law (guardianship, curatorship)
* Person under psychiatric care
* Person participating in another research project with an exclusion period still in progress,

Ages: 14 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Juvenile sex offenders
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
The feelings of patients who participated on a psychoeducation group | At the end of the 10 sessions (week 10) of the psychoeducation group
  One Guided Interview :
  The analysis of the interviews uses a phenomenological method aimed at bringing out data from the lived experience collected in the verbatims, each representing an aspect of the phenomenon studied.
  The raw data will be prepared in a word document. After a division into units of meaning and thematization by an inductive coding procedure using classificatory logic, the analysis consists of identifying the relevant elements in relation to the research question and in particular in relation to the chosen indicators. These different indicators will constitute an a priori analysis grid. They will be distributed in the different "boxes" previously established concerning the chosen indicators.
  Apart from these a priori indicators, concepts not planned in advance will be reported Patient's expectations before the group, description of the lived experience, emotions felt between two sessions, group description, patient's feed back after their participation.

SECONDARY OUTCOMES:
Socio-demographic data | At the end of the 10 sessions (week 10) of the psychoeducation group
  age and criminal records

CONTACTS AND LOCATIONS:
Overall Officials: celine BAIS, Ph, Study Director — University Hospital, Montpellier
Locations (1):
- UH MONTPELLIER - La Colombiere CRIAVS, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided